CLINICAL TRIAL: NCT01402830
Title: DPRESS Study. Case-control Study in Cancer Pain: Uncontrolled Pain as Depression Development Predictor in Oncologic Patients
Brief Title: Case-control Study- Cancer Pain: Uncontrolled Pain as Depression Development Predictor in Oncologic Patients (Fentanyl)
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag, S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR017656; FENPAI4055
Record Dates: First submitted 2011-07-25; First posted 2011-07-26 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: Cancer Pain
Keywords: cancer; depression; pain
MeSH Terms: conditions — Cancer Pain; Neoplasms; Depression; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- 001: Visual analogue scales (EVAs) This scale measures the pain intensity.
  Interventions: Other: Visual analogue scales (EVAs)

INTERVENTIONS:
Other: Visual analogue scales (EVAs) — This scale measures the pain intensity.

SUMMARY:
The purpose of this study is to evaluate the relationship between cancer pain and risk of depression among cancer patients.

DETAILED DESCRIPTION:
This is a retrospective observational and case-control multicenter study. The main objective of this study is determine the degree of association between cancer pain and depression by impact assessment of adequate control of pain associated with cancer risk depression in patients attending the Oncology Unit. The assessment of pain intensity will be performed by using visual analogue scales (EVAs) and verbal descriptive scales, as an observational study, not limit or modify the use of any drug. The patients included in this study have a medical history of cancer pain and mild depression (Beck = 8). The controls are patients with history of cancer pain and mild or absent depression (Beck = 7). n/a

ELIGIBILITY:
Inclusion Criteria:

* Patients =18 years old
* have medical data of = 3 months
* experience pain after cancer diagnosis and complete the Beck Depression Inventory (BDI)
* patients who give informed written consent
* patients with no mental or physical disorders that unable them to complete the BDI.

Exclusion Criteria:

* Patients with diagnosis of depression before cancer diagnosis
* patients with chronic pain prior to the diagnosis of cancer, and cancer disease has not changed its course
* patients with other previous mental disorders
* patients who do not give their informed written consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with cancer pain who experience depression and pain after cancer diagnosis
Sampling Method: Probability Sample
Enrollment: 271 (Actual)
Dates: Start 2007-11; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory | 3 months
Visual scales analog (EVAs) | 3 months

SECONDARY OUTCOMES:
Number of patients with cancer pain. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag S.A. (formerly Janssen Sp) Clinical Trial, Study Director — Janssen-Cilag, S.A.